CLINICAL TRIAL: NCT05430321
Title: The Effect of Facilitated Tucking After Vaginal Delivery on Late Preterm Stress, Comfort and Physiological Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Kilis 7 Aralik University (Other)
Responsible Party: Principal Investigator, SERAP ÖZDEMİR, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Istanbul
Record Dates: First submitted 2021-10-04; First posted 2022-06-24 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2022-06

CONDITIONS: Preterm Labor; Preterm Labor with Preterm Delivery in Third Trimester; Preterm Spontaneous Labor with Preterm Delivery
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Effect of facilitated tucking after preterm labor (Experimental): Implementation of facilitated tucking after preterm labor
  Interventions: Other: Assessment of physiological parameters; Other: Assessment of Stress; Other: Assessment of Comfort
- Supine position after preterm labor (No Intervention): Implementation of supine position after preterm labor

INTERVENTIONS:
Other: Assessment of physiological parameters — FT implementation begins 3 minutes before the procedures and 10 minutes continuous. After the end of the procedures further 3 minutes was given . Physiological parameters were simultaneously recorded on the registration form
  Arms: Effect of facilitated tucking after preterm labor
Other: Assessment of Stress — Newborn Stress Scale (NSS) was used end of the all procedures which means 13th minute.
  Arms: Effect of facilitated tucking after preterm labor
Other: Assessment of Comfort — Neonatal Comfort Behavior Scale (NCBS) was used end of the all procedures which means 13th minute.
  Arms: Effect of facilitated tucking after preterm labor

SUMMARY:
Objective: It is aimed to examine the effect of facilitated tucking after vaginal delivery on late preterm stress, comfort and physiological parameters.

Design: The study was designed randomized controlled study. Setting: The study was conducted spontaneous vaginal delivery of late preterm at State Hospital between January-June 2020.

Participants: In order to determine the sample size of the study, power analysis was performed using the G*Power (v3.1, 7) program, and a total of 60 preterm were sampled, facilitated tucking (n=30) and control group (n=30).

Methods: In the study, Newborn Information and Registration Form, Neonatal Comfort Behavior Scale (NCBS) and Newborn Stress Scale (NSS) were used. As for physiological parameters, for the temperature is used private digital thermometer, for the saturation and heart rate is used device preferred in hospital routine and lastly the respirator rate is clocked by nurses.

DETAILED DESCRIPTION:
Facilitated tucking (FT) is a procedure that kindly flexes the newborn by placing hands on the head and hips. There is no mentioned any risk about this implementation in the literature review. Its effects are that it improves the sleep quality of the newborn and stabilizes the physiological parameters helps to gain a sense of safety related to the position, support the motor development and protect the energy. Studies have shown that facilitated tucking is practiced many times, especially pain management; however, no study has been found examining how it affects stress and comfort of the preterm newborns first nursing care after delivery. Furthermore, vaginal delivery can be a cause of stress alone for all newborns. During these procedures, nursing practices are needed to relieve the stress and to provide comfort on the newborn. Therefore, it is aimed to examine the effect of facilitated tucking after vaginal delivery on late preterm stress, comfort and physiological parameters.

Material and Method: Power analysis for the present study was based on the study by a study which performed the study with at least 32, 30 preterm in each group (with 95% confidence interval and 5% alpha (two tailed)). Herein, the present study was performed with a total of 60 preterm corresponding to 30 preterm for each experimental group (It was assumed that could be lost cases during the study).Randomization was achieved by means of the computer program (https://www.randomizer.org) indicating the total number of preterm, groups and preterm groups and the preterm divided into control and experimental groups.

Experimental group: In order to eliminate the pain and stress that they experience during routine care after vaginal delivery to late preterm. FT implementation begins 3 minutes before the procedures and 10 minutes continuous. After the end of the procedures further 3 minutes was given. Physiological parameters were simultaneously recorded on the registration form. Neonatal Comfort Behavior Scale (NCBS) and Newborn Stress Scale (NSS) were used end of the all procedures which means 13th minute. While FT was implemented by researcher, postpartum care for newborn was performed and recorded by same nurse who is on shift. Evaluation of the scales was evaluated by the researcher and the nurse working in the hospital shift (with 5 years of neonatal experience) (Observer I-Observer II).

Control group: In this group was implemented of the hospital routine care (supine position). Physiological parameters were simultaneously recorded after the vaginal delivery. Neonatal Comfort Behavior Scale (NCBS) and Newborn Stress Scale (NSS) were used end of the all procedures which means 13th minute. Evaluation of the scales was evaluated by the researcher and the nurse working in the hospital shift (with 5 years of neonatal experience) (Observer I-Observer II).

ELIGIBILITY:
Inclusion Criteria:

* spontaneous vaginal delivery,
* Apgar score 1. min > 7
* between 35-36 (6/7) gestation weeks,
* without congenital anomaly or any syndrome,
* surgery is not needed,
* mechanical ventilation is not needed,
* accepted by parents.

Exclusion Criteria:

* in addition to the exact opposite of the items identified in the inclusion criteria, also cesarean, neonatal resuscitation is needed, newborn first vaccinations practices excluded.

Ages: 1 Hour to 2 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Sample characteristic | 13 minutes
  the characteristics of the preterm infants and their mothers in the groups.
Physiological parameter (Heart rate)-1 | 13 minutes
  the parameters (heart rate) of the groups were compared at hospitalization, 1st, 5th, 10th and 13th minutes.
Physiological parameter (oxygen saturation)-2 | 13 minutes
  the parameters (oxygen saturation) of the groups were compared at hospitalization, 1st, 5th, 10th and 13th minutes.
Physiological parameter (respiratory rate)-3 | 13 minutes
  It was stated that the parameters (respiratory rate) of the groups.
Neonatal Stress Scale scores | 13 minutes
  It was stated that the mean Neonatal Stress Scale scores between groups (min=3 max=11).
Newborn Comfort Behaviour Scale scores | 13 minutes
  It was determined that the mean Newborn Comfort Behaviour Scale scores between groups (min=6 max 30).
Physiological parameter (body temperature)-4 | 13 minutes
  It was observed that the parameters (body temperature).

CONTACTS AND LOCATIONS:
Overall Officials: Feyza Bulbul, PhD, Principal Investigator — Pediatric Nursing
Locations (1):
- Serap ÖZDEMİR, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Researchers would like to share all manuscript other colleges if this study is published.
Supporting Information: Study Protocol
Time Frame: 2 years
Access Criteria: If this study is published, than will share

REFERENCES:
- [Background] Hartley KA, Miller CS, Gephart SM. Facilitated tucking to reduce pain in neonates: evidence for best practice. Adv Neonatal Care. 2015 Jun;15(3):201-8. doi: 10.1097/ANC.0000000000000193. PMID 26002861
- [Background] Apaydin Cirik V, Efe E. The effect of expressed breast milk, swaddling and facilitated tucking methods in reducing the pain caused by orogastric tube insertion in preterm infants: A randomized controlled trial. Int J Nurs Stud. 2020 Apr;104:103532. doi: 10.1016/j.ijnurstu.2020.103532. Epub 2020 Jan 24. PMID 32062050
- [Background] Cignacco E, Axelin A, Stoffel L, Sellam G, Anand K, Engberg S. Facilitated tucking as a non-pharmacological intervention for neonatal pain relief: is it clinically feasible? Acta Paediatr. 2010 Dec;99(12):1763-5. doi: 10.1111/j.1651-2227.2010.01941.x. PMID 20618166
- [Background] Davari S, Borimnejad L, Khosravi S, Haghani H. The effect of the facilitated tucking position on pain intensity during heel stick blood sampling in premature infants: a surprising result. J Matern Fetal Neonatal Med. 2019 Oct;32(20):3427-3430. doi: 10.1080/14767058.2018.1465550. Epub 2018 Apr 26. PMID 29656669
- [Background] Gautheyrou L, Durand S, Jourdes E, De Jonckheere J, Combes C, Cambonie G. Facilitated tucking during early neonatologist-performed echocardiography in very preterm neonates. Acta Paediatr. 2018 Dec;107(12):2079-2085. doi: 10.1111/apa.14555. Epub 2018 Sep 21. PMID 30144169